CLINICAL TRIAL: NCT05523297
Title: Prospective, Multicenter, Active-control Randomized Trial Comparing 4-factor Prothrombin Complex Concentrate With Frozen Plasma in Bleeding Adult Cardiac Surgical Patients
Brief Title: Active-control Randomized Trial Comparing 4-factor Prothrombin Complex Concentrate With Frozen Plasma in Cardiac Surgery
Acronym: FARES-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEX-211
Record Dates: First submitted 2022-08-18; First posted 2022-08-31 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Bleeding Cardiac Surgery Patients
MeSH Terms: interventions — prothrombin complex concentrates

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Given the physical differences in the products and the emergency nature of the intervention, attending clinicians present during the infusion of the blood products/components were not blinded to the treatment. To minimize bias, treating clinicians were blinded to group assignments until immediately prior to IMP infusion. The sponsor and data management teams were also blinded to treatment group allocations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Octaplex (Experimental): Participants were administered Octaplex according to a recommended initial dose of 1,500 IU for patients weighing ≤60 kg and 2,000 IU for patients weighing >60 kg. A second dose of IMP could be administered if the patient continued to have at least moderate bleeding and suspected coagulation deficiency (e.g., INR ≥1.5) after completion of the first dose, up to the maximum allowable dose (3,000 IU if ≤60 kg or 4,000 IU if >60 kg).
  Octaplex: Prothrombin complex concentrate
  Interventions: Drug: Octaplex
- Frozen plasma (Active Comparator): Participants were administered FP according to a recommended initial dose of 3 U for patients weighing ≤60 kg and 4 U for patients weighing >60 kg. A second dose of IMP could be administered if the patient continued to have at least moderate bleeding and suspected coagulation deficiency (e.g., INR ≥1.5) after completion of the first dose, up to the maximum allowable dose (6 U if ≤60 kg or 8 U if >60 kg).
  Frozen Plasma Product, Human
  Interventions: Drug: Frozen Plasma Product, Human

INTERVENTIONS:
Drug: Octaplex — Prothrombin complex concentrate
  Arms: Octaplex
Drug: Frozen Plasma Product, Human — If additional treatment is required after the maximum dose of IMP is administered or the treatment period has elapsed, patients in both groups will receive frozen plasma
  Arms: Frozen plasma

SUMMARY:
This is a multicenter, active-control randomized, prospective, Phase 3 study in adult cardiac surgery patients. 420 patients were randomized at 12 hospitals.

DETAILED DESCRIPTION:
Patients were randomized to receive either 4-factor PCC (Octaplex) or frozen plasma (FP). The study compared the hemostatic treatment response to Octaplex versus FP, defined as effective if no additional systemic or surgical hemostatic intervention is required from 60 minutes to 24 hours after initiation of the first treatment dose. The study includes adult (≥18 years old) patients who underwent cardiac surgery with cardiopulmonary bypass (CPB) and required coagulation factor replacement due to bleeding post-CPB and after adequate reversal of heparin with protamine (as assessed by the surgical staff based on clinical and laboratory criteria) during surgery, and who have a known (e.g., as indicated by INR) or suspected coagulation factor deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years old) patients undergoing any index cardiac surgery employing CPB
2. Coagulation factor replacement with PCC or FP ordered in the operating room for:

   1. Management of bleeding, or
   2. Anticipated bleeding in a patient who has been on-pump for >2 hours or has undergone a complex procedure (e.g., aortocoronary bypass [ACB] plus aortic valve replacement)
3. Coagulation factor deficiency, either known to exist (e.g., as indicated by elevated EXTEM clotting time [CT] or INR) or suspected based on the clinical situation
4. Patients who have given written informed consent. In United States patients will provide informed consent prior to surgery. In Canada, informed consent will be obtained after surgery, in accordance with Article 3.7A of the 2018 Tri- Council Policy Statement on the Ethical Conduct for Research Involving Humans.

Exclusion Criteria:

1. Undergoing heart transplantation, insertion or removal of ventricular assist devices (not including intra-aortic balloon pump [IABP]) or repair of thoracoabdominal aneurysm
2. Critical state immediately before surgery with high probability of death within 24 hours of surgery (e.g., acute aortic dissection, cardiac arrest within 24 hours before surgery)
3. Severe right heart failure (clinical diagnosis ± echocardiography)
4. Known contraindications to heparin
5. PCC required for reversal of warfarin or direct oral anticoagulant (DOAC; dabigatran, rivaroxaban, apixaban or edoxaban) within 3 days prior to or during surgery
6. Known thromboembolic event (TEE) within 3 months prior to surgery
7. History of severe allergic reactions to PCC or FP
8. Individuals who have immunoglobulin A (IgA) deficiency with known antibodies against IgA
9. Refusal of allogeneic blood products
10. Known pregnancy
11. Currently enrolled in other interventional clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (2):
  - Duke University Health System, Durham, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
- Canada (11):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - University of British Columbia and Vancouver Coastal Health Authority, Vancouver, British Columbia
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Quebec Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karkouti K, Callum JL, Bartoszko J, Tanaka KA, Knaub S, Brar S, Ghadimi K, Rochon A, Mullane D, Couture EJ, Lin Y, Harle C, Zeller M, Tran DTT, Solomon C, Rao V, Law M, Butt AL, Chen EP, Martins MR, Saha T, Shih AW, Vezina MC, Moussa F, Pereira Cezar Zamper R, Syed S, Buyukdere H, Werner S, Grewal D, Wong D, Vandyck KB, Tanzola R, Hughes B, Royer O, Wong S, Levy JH; FARES-II Study Group. Prothrombin Complex Concentrate vs Frozen Plasma for Coagulopathic Bleeding in Cardiac Surgery: The FARES-II Multicenter Randomized Clinical Trial. JAMA. 2025 May 27;333(20):1781-1792. doi: 10.1001/jama.2025.3501. PMID 40156829
- [Derived] Karkouti K, Callum J, Bartoszko J, Solomon C, Knaub S, Levy JH, Tanaka KA; FARES-II Study Group. Protocol for a phase 3, randomised, active-control study of four-factor prothrombin complex concentrate versus frozen plasma in bleeding adult cardiac surgery patients requiring coagulation factor replacement: the LEX-211 (FARES-II) trial. BMJ Open. 2024 Aug 21;14(8):e091381. doi: 10.1136/bmjopen-2024-091381. PMID 39174056

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 10 Canadian sites and 2 US sites. The first participant was enrolled in November 2022 and the last patient completed the study in June 2024.
Pre-assignment Details: Of 538 enrolled participants, 420 met the inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | Octaplex | Frozen Plasma
Started | 213 | 207
Per-protocol Population (PP) | 209 | 200
Completed | 204 | 198
Not Completed | 9 | 9
Not completed — Death | 7 | 8
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Octaplex | Frozen Plasma | Total
Number analyzed (Participants) | 213 | 207 | 420
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.97 (13.596) | 61.68 (14.002) | 62.84 (13.829)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 55 | 111
  Male | 157 | 152 | 309
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 132 | 132 | 264
  Unknown or Not Reported | 79 | 73 | 152
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 20 | 21 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 138 | 137 | 275
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 49 | 45 | 94
Body Height [Mean (Standard Deviation); unit: centimeter (cm)] | 171.03 (10.082) | 171.83 (10.565) | 171.42 (10.318)
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 84.63 (19.344) | 83.62 (19.520) | 84.13 (19.414)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m²)] | 28.88 (5.986) | 28.20 (5.403) | 28.55 (5.710)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Requiring Additional Hemostatic Intervention
Description: Defined as 'effective' if no additional hemostatic intervention, such as administration of any systemic hemostatic agents (including platelets, cryoprecipitate, fibrinogen concentrate, activated recombinant factor VII [rFVIIa], other coagulation factor products or a second dose of IMP) or any hemostatic interventions (including surgical re-opening for bleeding) is required from 60 minutes to 24 hours after initiation of the first dose of IMP.
Time Frame: 60 minutes to 24 hours after first dose of IMP
Measure: Count of Participants; unit: Participants
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 207
Participants
  Effective | 166 | 125
  Ineffective | 47 | 82
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; Test type: Non-Inferiority — The test for non-inferiority was one-sided Farrington-Manning score test with non-inferiority margin 10% at a significance level of 2.5%. If the 95% CI for treatment effect not only lay above -10% (the non-inferiority margin) but also above 0, then there was evidence of superiority; p < 0.0001, Two-sided Farrington-Manning score test; percent difference = 17.55, 95% CI 2-sided [8.7 to 26.4] — Difference between Octaplex and FP arms for effectiveness

2. Secondary Outcome: Comparison of Global Hemostatic Response Based on Requirement of Additional Hemostatic Intervention and Decreased Hemoglobin Levels
Description: Defined as 'positive' if no additional hemostatic intervention is required and hemoglobin levels decrease by <30% (after accounting for red cell transfusions) from 60 minutes to 24 hours after initiation of the first dose of IMP.
Time Frame: 60 minutes to 24 hours after first dose of IMP
Population: Data were not available for 2 patients in the FP group due to missing hemoglobin values.
Measure: Count of Participants; unit: Participants
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 205
Participants
  Negative | 56 | 83
  Positive | 157 | 122
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; Test type: Other; p = 0.0022, Regression, Logistic; Odds Ratio (OR) = 1.91, 95% CI 2-sided [1.26 to 2.88]

3. Secondary Outcome: Compare the Amount of Chest Tube Drainage Between the Octaplex and FP Groups.
Time Frame: 12 and 24 hours after chest closure
Measure: Mean (Standard Deviation); unit: Milliliters (mL)
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 207
Milliliters (mL)
  12 hours after chest closure | 471.20 (358.32) | 641.90 (465.17)
  24 hours after chest closure | 690.90 (465.62) | 922.90 (631.90)
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; 12 hours after chest closure; Test type: Other; p < 0.0001, ANOVA; Least Squares Mean Difference = -170.73, 95% CI 2-sided [-250.24 to -91.22]
Statistical Analysis 2: Comparison: Octaplex vs Frozen Plasma; 24 hours after chest closure; Test type: Other; p < 0.0001, ANOVA; Least Squares Mean Difference = -231.92, 95% CI 2-sided [-338.17 to -125.67]

4. Secondary Outcome: Compare the Incidence of Severe to Massive Bleeding Between the Octaplex and FP Groups Using a Modification of the Universal Definition of Perioperative Bleeding (UDPB).
Description: Yes or no refers to whether severe to massive bleeding was present.
Time Frame: 24 hours after surgery start, after the end of CPB and after IMP initiation
Measure: Count of Participants; unit: Participants
Groups:
- Octaplex: Participants received up to 2 Octaplex infusions intravenously within the first 24 hours. The recommended initial dose for Octaplex was 1,500 IU for patients weighing ≤60 kg and 2,000 IU for patients weighing >60 kg. A second dose of IMP could be administered if the patient continued to have at least moderate bleeding and suspected coagulation deficiency (e.g., INR ≥1.5) after completion of the first dose, up to the maximum allowable dose (3,000 IU if ≤60 kg or 4,000 IU if >60 kg).
  Beyond 24 hours after initiation of the first dose, frozen plasma was administered if further coagulation factor replacement therapy was ordered.
  Octaplex: Prothrombin complex concentrate
- Frozen Plasma: Participants were administered FP according to a recommended initial dose of 3 U for patients weighing ≤60 kg and 4 U for patients weighing >60 kg. A second dose of IMP could be administered if the patient continued to have at least moderate bleeding and suspected coagulation deficiency (e.g., INR ≥1.5) after completion of the first dose, up to the maximum allowable dose (6 U if ≤60 kg or 8 U if >60 kg).
  Frozen Plasma Product, Human: If additional coagulation factor replacement therapy was required after the maximum dose of IMP was administered or the 24-hour treatment period had elapsed, patients in both groups received frozen plasma.
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 207
Participants
  Within 24 hours after IMP start: No | 183 | 136
  Within 24 hours after IMP start: Yes | 30 | 71
  Within 24 hours after surgery start: No | 176 | 129
  Within 24 hours after surgery start: Yes | 37 | 78
  Within 24 hours after CBP end: No | 183 | 136
  Within 24 hours after CBP end: Yes | 30 | 71
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; Within 24 hours after IMP start; Test type: Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.19, 95% CI 2-sided [1.97 to 5.15]
Statistical Analysis 2: Comparison: Octaplex vs Frozen Plasma; Within 24 hours after surgery start; Test type: Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.88, 95% CI 2-sided [1.83 to 4.52]
Statistical Analysis 3: Comparison: Octaplex vs Frozen Plasma; Within 24 hours after CPB end; Test type: Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.19, 95% CI 2-sided [1.97 to 5.15]

5. Secondary Outcome: Compare Efficacy in Terms of the Mean Number of Total Allogeneic Blood Products (ABPs) (IMP and Non-IMP) Transfused Between the Octaplex and FP Groups.
Time Frame: First 24 hours after the end of CPB
Measure: Mean (Standard Deviation); unit: total ABPs
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 207
total ABPs | 6.61 (6.95) | 13.79 (11.42)
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; Test type: Other; p < 0.0001, Counting regression; Mean ratio = 0.48, 95% CI 2-sided [0.41 to 0.57]

6. Secondary Outcome: Compare Efficacy in Terms of the Mean Number of Total Non-IMP Allogeneic Blood Products Transfused Between the Octaplex and FP Groups.
Time Frame: First 24 hours after the end of CPB
Measure: Mean (Standard Deviation); unit: total non-IMP ABPs
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 207
total non-IMP ABPs | 6.61 (6.95) | 9.33 (10.64)
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; Test type: Other; p = 0.0015, Counting regression; Mean ratio = 0.71, 95% CI 2-sided [0.57 to 0.88]

7. Secondary Outcome: Compare Efficacy in Terms of the Mean Number of Total Non-IMP Allogeneic Blood Components Transfused Between the Octaplex and FP Groups.
Time Frame: First 24 hours and 7 days after IMP initiation
Measure: Mean (Standard Deviation); unit: Total non-IMP ABPs
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 207
Total non-IMP ABPs
  During the first 24 hours after IMP start | 4.14 (6.25) | 6.73 (10.14)
  During the first 7 days after IMP start | 5.20 (8.43) | 8.87 (16.04)
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; During the first 24 hours after IMP start; Test type: Other; p = 0.0010, Counting regression; Mean ratio = 0.61, 95% CI 2-sided [0.46 to 0.82]
Statistical Analysis 2: Comparison: Octaplex vs Frozen Plasma; During the first 7 days after IMP start; Test type: Other; p < 0.0001, Counting regression; Mean ratio = 0.59, 95% CI 2-sided [0.45 to 0.76]

8. Secondary Outcome: Compare Mean Number of Individual Allogeneic Blood Components Transfused Between the Octaplex and FP Groups.
Time Frame: 24 hours and 7 days after start of surgery, and after the end of CPB and after IMP initiation
Measure: Mean (Standard Deviation); unit: ABPs
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 207
ABPs
  FP including IMP (During the first 24 hours after IMP start) | 0.19 (1.12) | 4.70 (2.47)
  FP excluding IMP (During the first 24 hours after IMP start) | 0.19 (1.12) | 0.23 (1.63)
  RBCs (During the first 24 hours after IMP start) | 1.05 (1.72) | 2.02 (2.58)
  Platelets (During the first 24 hours after IMP start) | 2.89 (4.50) | 4.48 (6.80)
  Cryoprecipitate (During the first 24 hours after IMP start) | 0.08 (0.42) | 0.14 (0.61)
  FP including IMP (During the first 7 days after IMP start) | 0.23 (1.273) | 7.25 (34.818)
  FP excluding IMP (During the first 7 days after IMP start) | 0.23 (1.273) | 2.78 (34.792)
  Red blood cells (During the first 7 days after IMP start) | 1.7 (2.378) | 2.9 (3.466)
  Platelets (During the first 7 days after IMP start) | 3.27 (5.827) | 5.6 (11.530)
  Cryoprecipitate (During the first 7 days after IMP start) | 0.08 (0.421) | 0.16 (0.765)
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; FP including IMP (During the first 24 hours after IMP start); Test type: Other; p < 0.0001, Negative binomial regression; Mean ratio = 0.04, 95% CI 2-sided [0.03 to 0.06]
Statistical Analysis 2: Comparison: Octaplex vs Frozen Plasma; FP excluding IMP (During the first 24 hours after IMP start); Test type: Other; p = 0.8522, Negative binomial regression; Mean ratio = 0.85, 95% CI 2-sided [0.15 to 4.82]
Statistical Analysis 3: Comparison: Octaplex vs Frozen Plasma; RBCs (During the first 24 hours after IMP start); Test type: Other; p < 0.0001, Negative binomial regression; Mean ratio = 0.52, 95% CI 2-sided [0.40 to 0.68]
Statistical Analysis 4: Comparison: Octaplex vs Frozen Plasma; Platelets (During the first 24 hours after IMP start); Test type: Other; p = 0.0169, Negative binomial regression; Mean ratio = 0.65, 95% CI 2-sided [0.45 to 0.92]
Statistical Analysis 5: Comparison: Octaplex vs Frozen Plasma; Cryoprecipitate (During the first 24 hours after IMP start); Test type: Other; p = 0.3288, Negative binomial regression; Mean ratio = 0.57, 95% CI 2-sided [0.18 to 1.76]
Statistical Analysis 6: Comparison: Octaplex vs Frozen Plasma; FP including IMP (During the first 7 days after IMP start); Test type: Other; p < 0.0001, Negative binomial regression; Mean ratio = 0.05, 95% CI 2-sided [0.04 to 0.06]
Statistical Analysis 7: Comparison: Octaplex vs Frozen Plasma; FP excluding IMP (During the first 7 days after IMP start); Test type: Other; p = 0.5439, Negative binomial regression; Mean ratio = 0.63, 95% CI 2-sided [0.14 to 2.84]
Statistical Analysis 8: Comparison: Octaplex vs Frozen Plasma; Red blood cells (During the first 7 days after IMP start); Test type: Other; p < 0.0001, Negative binomial regression; Mean ratio = 0.59, 95% CI 2-sided [0.47 to 0.74]
Statistical Analysis 9: Comparison: Octaplex vs Frozen Plasma; Platelets (During the first 7 days after IMP start); Test type: Other; p = 0.0042, Negative binomial regression; Mean ratio = 0.58, 95% CI 2-sided [0.40 to 0.84]
Statistical Analysis 10: Comparison: Octaplex vs Frozen Plasma; Cryoprecipitate (During the first 7 days after IMP start); Test type: Other; p = 0.2241, Negative binomial regression; Mean ratio = 0.49, 95% CI 2-sided [0.15 to 1.56]

9. Secondary Outcome: Compare Efficacy in Terms of the Incidence of Transfusion of Individual Allogeneic Blood Components Transfused Between the Octaplex and FP Groups.
Time Frame: 24 hours and 7 days after start of surgery and after the end of CPB and after IMP initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 207
Participants
  FP excluding IMP (Within 24 hours after IMP start): No | 205 | 200
  FP excluding IMP (Within 24 hours after IMP start): Yes | 8 | 7
  RBCs (Within 24 hours after IMP start): No | 116 | 75
  RBCs (Within 24 hours after IMP start): Yes | 97 | 132
  Platelets (Within 24 hours after IMP start): No | 116 | 99
  Platelets (Within 24 hours after IMP start): Yes | 97 | 108
  Cryoprecipitate (Within 24 hours after IMP start): No | 204 | 195
  Cryoprecipitate (Within 24 hours after IMP start): Yes | 9 | 12
  Any individual ABP (Within 24 hours after IMP start): No | 82 | 56
  Any individual ABP (Within 24 hours after IMP start): Yes | 131 | 151
  FP excluding IMP (Within 7 days after IMP start): No | 205 | 195
  FP excluding IMP (Within 7 days after IMP start): Yes | 8 | 12
  RBCs (Within 7 days after IMP start): No | 82 | 53
  RBCs (Within 7 days after IMP start): Yes | 131 | 154
  Platelets (Within 7 days after IMP start): No | 112 | 97
  Platelets (Within 7 days after IMP start): Yes | 101 | 110
  Cryoprecipitate (Within 7 days after IMP start): No | 204 | 195
  Cryoprecipitate (Within 7 days after IMP start): Yes | 9 | 12
  Any individual ABP (Within 7 days after IMP start): No | 58 | 40
  Any individual ABP (Within 7 days after IMP start): Yes | 155 | 167
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; FP excluding IMP (Within 24 hours after IMP start); Test type: Other; p = 0.8364, Regression, Logistic; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.32 to 2.52]
Statistical Analysis 2: Comparison: Octaplex vs Frozen Plasma; RBCs (Within 24 hours after IMP start); Test type: Other; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 2.11, 95% CI 2-sided [1.42 to 3.11]
Statistical Analysis 3: Comparison: Octaplex vs Frozen Plasma; Platelets (Within 24 hours after IMP start); Test type: Other; p = 0.1742, Regression, Logistic; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.89 to 1.91]
Statistical Analysis 4: Comparison: Octaplex vs Frozen Plasma; Cryoprecipitate (Within 24 hours after IMP start); Test type: Other; p = 0.4618, Regression, Logistic; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.58 to 3.38]
Statistical Analysis 5: Comparison: Octaplex vs Frozen Plasma; Any individual ABP (Within 24 hours after IMP start); Test type: Other; p = 0.0129, Regression, Logistic; Odds Ratio (OR) = 1.69, 95% CI 2-sided [1.12 to 2.55]
Statistical Analysis 6: Comparison: Octaplex vs Frozen Plasma; FP excluding IMP (Within 7 days after IMP start); Test type: Other; p = 0.3297, Regression, Logistic; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.63 to 3.94]
Statistical Analysis 7: Comparison: Octaplex vs Frozen Plasma; RBCs (Within 7 days after IMP start); Test type: Other; p = 0.0049, Regression, Logistic; Odds Ratio (OR) = 1.82, 95% CI 2-sided [1.20 to 2.76]
Statistical Analysis 8: Comparison: Octaplex vs Frozen Plasma; Platelets (Within 7 days after IMP start); Test type: Other; p = 0.2417, Regression, Logistic; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.86 to 1.84]
Statistical Analysis 9: Comparison: Octaplex vs Frozen Plasma; Cryoprecipitate (Within 7 days after IMP start); Test type: Other; p = 0.4618, Regression, Logistic; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.58 to 3.38]
Statistical Analysis 10: Comparison: Octaplex vs Frozen Plasma; Any individual ABP (Within 7 days after IMP start); Test type: Other; p = 0.0564, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.99 to 2.47]

10. Secondary Outcome: Compare Incidence of Administration of Non-IMP Coagulation Factor Products Between Octaplex and FP Groups
Time Frame: 24 hours and 7 days after the start of surgery, after the end of CPB and after IMP initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 207
Participants
  Fibrinogen concentrate (Within 24 hours after IMP start): No | 167 | 159
  Fibrinogen concentrate (Within 24 hours after IMP start): Yes | 46 | 48
  rFVIIa (Within 24 hours after IMP start): No | 211 | 197
  rFVIIa (Within 24 hours after IMP start): Yes | 2 | 10
  PCC excluding IMP (Within 24 hours after IMP start): No | 212 | 190
  PCC excluding IMP (Within 24 hours after IMP start): Yes | 1 | 17
  Any coagulation factor product (Within 24 hours after IMP start): No | 164 | 148
  Any coagulation factor product (Within 24 hours after IMP start): Yes | 49 | 59
  Fibrinogen concentrate (Within 7 days after IMP start): No | 167 | 156
  Fibrinogen concentrate (Within 7 days after IMP start): Yes | 46 | 51
  rFVIIa (Within 7 days after IMP start): No | 211 | 197
  rFVIIa (Within 7 days after IMP start): Yes | 2 | 10
  PCC excluding IMP (Within 7 days after IMP start): No | 212 | 190
  PCC excluding IMP (Within 7 days after IMP start): Yes | 1 | 17
  Any coagulation factor product (Within 7 days after IMP start): No | 164 | 145
  Any coagulation factor product (Within 7 days after IMP start): Yes | 49 | 62
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; Fibrinogen concentrate (Within 24 hours after IMP start); Test type: Other; p = 0.6956, Regression, Logistic; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.69 to 1.73]
Statistical Analysis 2: Comparison: Octaplex vs Frozen Plasma; Test type: Other; p = 0.0317, Regression, Logistic; Odds Ratio (OR) = 5.337, 95% CI 2-sided [1.12 to 50.70]
Statistical Analysis 3: Comparison: Octaplex vs Frozen Plasma; PCC excluding IMP (Within 24 hours after IMP start); Test type: Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 18.880, 95% CI 2-sided [2.90 to 796.37]
Statistical Analysis 4: Comparison: Octaplex vs Frozen Plasma; Any coagulation factor product (Within 24 hours after IMP start); Test type: Other; p = 0.1981, Regression, Logistic; Odds Ratio (OR) = 1.334, 95% CI 2-sided [0.86 to 2.07]
Statistical Analysis 5: Comparison: Octaplex vs Frozen Plasma; Fibrinogen concentrate (Within 7 days after IMP start); Test type: Other; p = 0.4599, Regression, Logistic; Odds Ratio (OR) = 1.187, 95% CI 2-sided [0.75 to 1.87]
Statistical Analysis 6: Comparison: Octaplex vs Frozen Plasma; rFVIIa (Within 7 days after IMP start); Test type: Other; p = 0.0317, Regression, Logistic; Odds Ratio (OR) = 5.337, 95% CI 2-sided [1.12 to 50.70]
Statistical Analysis 7: Comparison: Octaplex vs Frozen Plasma; PCC excluding IMP (Within 7 days after IMP start); Test type: Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 18.880, 95% CI 2-sided [2.90 to 796.37]
Statistical Analysis 8: Comparison: Octaplex vs Frozen Plasma; Any coagulation factor product (Within 7 days after IMP start); Test type: Other; p = 0.1073, Regression, Logistic; Odds Ratio (OR) = 1.431, 95% CI 2-sided [0.93 to 2.21]

11. Secondary Outcome: Compare Incidence of Intracerebral Hemorrhage Between the Octaplex and FP Groups
Time Frame: 24 hours after start of surgery, after the end of CPB and after IMP initiation
Measure: Number; unit: participants
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 207
participants
  24 hours after start of surgery | 0 | 0
  After the end of CPB | 0 | 0
  After IMP initiation | 0 | 0

12. Secondary Outcome: Compare Incidence of Gastrointestinal Hemorrhage Between Octaplex and FP Groups
Time Frame: 24 hours after start of surgery, after the end of CPB and after IMP initiation
Measure: Number; unit: participants
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 207
participants
  24 hours after start of surgery | 0 | 0
  After the end of CPB | 0 | 0
  After IMP initiation | 0 | 0

13. Secondary Outcome: Compare Incidence of Surgical Re-exploration Between Octaplex and FP Groups
Time Frame: 24 hours after start of surgery, after the end of CPB and after IMP initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 207
Participants
  Within 24 hours after surgery start: No | 200 | 189
  Within 24 hours after surgery start: Yes | 13 | 18
  Within 24 hours after CPB end: No | 199 | 187
  Within 24 hours after CPB end: Yes | 14 | 20
  Within 24 hours after IMP start: No | 199 | 187
  Within 24 hours after IMP start: Yes | 14 | 20
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; Within 24 hours after CPB end; Test type: Other; p = 0.3782, Regression, Logistic; Odds Ratio (OR) = 1.435, 95% CI 2-sided [0.6429 to 3.2013]
Statistical Analysis 2: Comparison: Octaplex vs Frozen Plasma; Within 24 hours after IMP start; Test type: Other; p = 0.3782, Regression, Logistic; Odds Ratio (OR) = 1.435, 95% CI 2-sided [0.6429 to 3.2013]
Statistical Analysis 3: Comparison: Octaplex vs Frozen Plasma; Within 24 hours after surgery start; Test type: Other; p = 0.4899, Regression, Logistic; Odds Ratio (OR) = 1.332, 95% CI 2-sided [0.5902 to 3.0062]

14. Secondary Outcome: Comparison of the Effect of Octaplex Versus FP Administration on the Change in International Normalised Ratio (INR) Before and After Therapy Administration.
Description: The international normalized ratio (INR) is a standardized measure of prothrombin time (PT), ensuring consistency in results across different laboratories. The normal range for INR is around 0.8 to 1.2. Higher INR values indicate a slower clotting time and are associated with bleeding. Effective procoagulant therapy can reduce/normalize the INR.
  INR reduction was considered successful if the magnitude of the reduction was >1.0 or the post-treatment level dropped below 1.5 (INR >1.5 indicates that one or more coagulation factor levels are below the 30% critical threshold)
Time Frame: Within 30 minutes before to 60 minutes after the initiation of IMP administration.
Population: The analysis of absolute change included all patients who had INR data available at both pre- and post-IMP time points.
Measure: Mean (Standard Deviation); unit: international normalised ratio (INR)
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 200 | 193
international normalised ratio (INR) | -0.9 (0.76) | -0.7 (0.91)
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; Test type: Other; p = 0.0081, ANOVA; Least Squares Mean Difference = -0.15, 95% CI 2-sided [-0.26 to -0.04]

15. Secondary Outcome: Comparison of the Effect of Octaplex Versus FP Administration on the Change in Prothrombin Time (PT)
Description: The prothrombin time (PT) measures the time it takes for clotting to occur, primarily assessing the extrinsic pathway of the coagulation cascade. Normal PT values range from 9 to 13 seconds. Higher PT values indicate a prolonged clotting time, suggesting potential issues with clotting factors such as fibrinogen, factors V, VII, and X and prothrombin, and are associated with bleeding. Effective procoagulant therapy can reduce/normalize the PT.
Time Frame: Within 75 minutes before to within 75 minutes after the initiation of IMP administration
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 9 | 1
seconds | -10.3 (20.90) | -0.7 (NA) — SD not available (n=1).
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; Test type: Other; p = 0.6735, ANOVA; Least Squares Mean Difference = -9.63, 95% CI 2-sided [-60.45 to 41.18]

16. Secondary Outcome: Comparison of the Effect of Octaplex Versus FP Administration on the Change in Activated Partial Thromboplastin Time (aPTT)
Description: Activated partial thromboplastin time (aPTT) is a standard laboratory test that measures how long it takes (in seconds) for clotting to occur (in the presence of an activator). It evaluates the intrinsic and common pathways of the coagulation cascade, assessing factors such as VIII, IX, XI, and XII, as well as fibrinogen. Prolonged aPTT may signify deficiencies in these clotting factors and is associated with bleeding. Effective procoagulant therapy can shorten/normalize the aPTT.
Time Frame: Within 75 minutes before to within 75 minutes after the initiation of IMP administration
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 4 | 1
seconds | -63.5 (121.47) | -45.6 (NA) — SD not available (n=1).
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; Test type: Other; p = 0.9033, ANOVA; Least Squares Mean Difference = -17.93, 95% CI 2-sided [-450.13 to 414.28]

17. Secondary Outcome: Comparison of the Effect of Octaplex Versus FP Administration on the Change in Fibrinogen Activity
Time Frame: Within 75 minutes before to within 75 minutes after the initiation of IMP administration
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 4 | 2
grams per liter (g/L) | 0.1 (0.07) | 0.5 (0.57)
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; Test type: Other; p = 0.1808, ANOVA; Least Squares Mean Difference = -0.41, 95% CI 2-sided [-1.10 to 0.29]

18. Secondary Outcome: Comparison of the Effect of Octaplex Versus FP Administration on the Change in ROTEM EXTEM CT
Description: A rotational thromboelastometry (ROTEM; Werfen) device can be used at the bedside to rapidly assess the patient's coagulation status. Different viscoelastic tests can be performed to assess the dynamics of clot formation and lysis. Specifically, the EXTEM test is activated with tissue factor and evaluates the extrinsic coagulation pathway, with clotting time (CT) providing a measure (in seconds) of how quickly a clot starts forming. Prolonged EXTEM CT is associated with bleeding. Effective procoagulant therapy can reduce/normalize the EXTEM CT.
Time Frame: Within 75 minutes before to within 75 minutes after the initiation of IMP administration
Population: Few data were available as ROTEM measurements were not mandated by the study protocol.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 11 | 15
seconds | -21.5 (18.00) | -21.7 (18.65)
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; Test type: Other; p = 0.9698, ANOVA; Least Squares Mean Difference = 0.28, 95% CI 2-sided [-14.78 to 15.34]

19. Secondary Outcome: Comparison of the Effect of Octaplex Versus FP Administration on the Change in ROTEM EXTEM MCF
Description: A rotational thromboelastometry (ROTEM; Werfen) device can be used at the bedside to rapidly assess the patient's coagulation status. Different viscoelastic tests can be performed to assess the dynamics of clot formation and lysis. Specifically, the EXTEM test is activated with tissue factor and evaluates the extrinsic coagulation pathway, with maximum clot firmness (MCF) providing a measure (in mm) of the strength of the clot. Reduced EXTEM MCF is associated with bleeding. Effective procoagulant therapy can increase/normalize the EXTEM MCF.
Time Frame: Within 75 minutes before to within 75 minutes after the initiation of IMP administration
Population: Few data were available as ROTEM measurements were not mandated by the study protocol.
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 11 | 15
Millimeters (mm) | 3.6 (4.95) | 6.7 (9.54)
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; Test type: Other; p = 0.3363, ANOVA; Least Squares Mean Difference = -3.10, 95% CI 2-sided [-9.61 to 3.42]

20. Secondary Outcome: Comparison of the Effect of Octaplex Versus FP Administration on the Change in ROTEM FIBTEM MCF
Description: A rotational thromboelastometry (ROTEM; Werfen) device can be used at the bedside to rapidly assess the patient's coagulation status. Different viscoelastic tests can be performed to assess the dynamics of clot formation and lysis. Specifically, the FIBTEM test evaluates fibrin-based clotting - it is extrinsically activated with tissue factor and additionally incorporates an inhibitor to eliminate the contribution of platelets to clotting. Maximum clot firmness (MCF) in the FIBTEM test provides a measure (in mm) of the strength of the fibrin-based clot. Reduced FIBTEM MCF is associated with bleeding. Effective procoagulant therapy to restore fibrinogen can increase/normalize the FIBTEM MCF.
Time Frame: Within 75 minutes before to within 75 minutes after the initiation of IMP administration
Population: Few data were available as ROTEM measurements were not mandated by the study protocol.
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 11 | 15
Millimeters (mm) | 3.8 (2.75) | 1.4 (13.78)
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; Test type: Other; p = 0.5736, ANOVA; Least Squares Mean Difference = 2.42, 95% CI 2-sided [-6.33 to 11.16]

21. Secondary Outcome: Comparison of the Effect of Octaplex Versus FP Administration on the Change in Platelet Count Measured by Plateletworks
Time Frame: Within 75 minutes before to within 75 minutes after the initiation of IMP administration
Population: The analysis of absolute change included all patients who had coagulation parameter data available at both pre- and post-IMP time points.
Measure: Mean (Standard Deviation); unit: 10^9 platelets/L
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 15 | 14
10^9 platelets/L | -2.3 (22.97) | 10.9 (38.29)
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; Test type: Other; p = 0.2667, ANOVA; Least Squares Mean Difference = -13.19, 95% CI 2-sided [-37.05 to 10.67]

22. Secondary Outcome: Comparison of the Effect of Octaplex Versus FP Administration on the Change in Platelet Function Measured by Plateletworks
Description: The Plateletworks device (Helena Laboratories) enables rapid bedside screening of platelet function. The system uses an impedance cell counter and Plateletworks reagent tubes to evaluate platelet function and monitor treatment effects. By comparing a baseline total platelet count against the platelet count measured in the presence of an agonist used to stimulate platelet aggregation (ADP, collagen, or arachidonic acid), the tests determine the percent aggregation or inhibition of functional platelets. Manufacturer reference ranges, determined by testing blood samples from healthy volunteers, are 86-100% for ADP, 70-100% for collagen, and 60-100% for arachidonic acid. Values within these ranges indicate 'normal (positive)' platelet aggregation, which is important for clotting; lower values may be considered 'abnormal (negative)' and reflective of platelet inhibition. The manufacturer advises each laboratory to establish their own reference ranges for their patient population.
Time Frame: Within 75 minutes before to within 75 minutes after the initiation of IMP administration
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 10 | 13
percentage | -5.9 (10.34) | -18.2 (17.72)
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; Test type: Other; p = 0.0658, ANOVA; Least Squares Mean Difference = 12.25, 95% CI 2-sided [-0.87 to 25.38]

23. Secondary Outcome: Comparison of Total Time Elapsed From Initiation of the First Dose of IMP to Arrival Into the ICU Between the Octaplex and FP Groups.
Time Frame: From initiation of IMP to arrival at ICU room (within 24 hours)
Population: 37 patients were excluded from the analysis population. 27 (12 in the Octaplex group, 25 in the FP group) who were already in the ICU when the first dose of IMP was initiated, 5 patients (2 in the Octaplex group, 3 in the FP group) for whom the time intervals could not be calculated due to incomplete date/time of arrival at ICU, and 1 patient (FP group) who was not in the ICU, therefore the time interval could not be calculated.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 199 | 178
hours | 1.0 [0.6 to 1.7] | 1.2 [0.7 to 2.0]
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; Test type: Other; p = 0.0726, ANOVA; Least Squares Mean Difference = -0.19, 95% CI 2-sided [-0.40 to 0.02]

24. Secondary Outcome: Comparison of Incidence of Serious Treatment-emergent Adverse Events Between Octaplex and FP Groups
Time Frame: From the beginning of surgery up to postoperative day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 207
Participants | 77 | 98

25. Secondary Outcome: Comparison of the Duration of Mechanical Ventilation Between Octaplex and FP Groups
Time Frame: From the beginning of surgery up to postoperative day 30
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 207
days | 1.0 [1 to 2] | 1.0 [1 to 2]

26. Secondary Outcome: Comparison of the Duration of ICU Stay Between Octaplex and FP Groups
Time Frame: From the beginning of surgery up to postoperative day 30
Population: Three patients in the FP group were excluded from this analysis due to missing dates of ICU stays
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 204
days | 4 [2 to 6] | 4 [2 to 7]

27. Secondary Outcome: Comparison of the Duration of Hospitalization Between Octaplex and FP Groups
Time Frame: From the beginning of surgery up to postoperative day 30
Population: One patient in the FP group was excluded from analysis due to missing data
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 206
days | 8 [7 to 12] | 9 [7 to 13]

28. Secondary Outcome: Comparison of the Incidence of Death Between Octaplex and FP Groups
Time Frame: Up to 30 days after the end of CPB
Measure: Count of Participants; unit: Participants
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 207
Participants | 7 | 8
Statistical Analysis 1: Comparison: Octaplex vs Frozen Plasma; Test type: Other; p = 0.7497, Regression, Logistic; Odds Ratio (OR) = 1.183, 95% CI 2-sided [0.4211 to 3.3235]

29. Secondary Outcome: Comparison of the Number of Days Alive and Out of Hospital Between Octaplex and FP Groups
Time Frame: From the beginning of surgery up to postoperative day 30
Population: One participant is excluded from analysis due to missing start/end date of hospitalization.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Octaplex | Frozen Plasma
Number analyzed (Participants) | 213 | 206
days | 21.0 [17.0 to 23.0] | 21.0 [16.0 to 23.0]

ADVERSE EVENTS:
Time Frame: From beginning of surgery to 30 days after surgery start
Arm/Group | Octaplex | Frozen Plasma
All-Cause Mortality (participants affected / at risk) | 7/213 | 8/207
Serious Adverse Events (participants affected / at risk) | 77/213 | 98/207
Other Adverse Events (participants affected / at risk) | 206/213 | 201/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octaplex (N=213) | Frozen Plasma (N=207)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Gall bladder abscess (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Graft infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia escherichia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Post procedural pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1)
Prosthetic valve endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 4 (4)
Septic shock (Infections and infestations) | 4 (4) | 2 (2)
Staphylococcal bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Stenotrophomonas bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Stenotrophomonas maltophilia pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypervolemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 5 (5)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Ischemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 4 (4)
Acute right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 7 (7) | 8 (10)
Atrial flutter (Cardiac disorders) | 3 (3) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 9 (9) | 3 (3)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 2 (2) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 5 (5)
Cardiac tamponade (Cardiac disorders) | 8 (8) | 5 (5)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 3 (3) | 8 (8)
Carditis (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Intrapericardial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Low cardiac output syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Nodal rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 3 (3)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 3 (3)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 2 (2)
Distributive shock (Vascular disorders) | 2 (2) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (1) | 1 (1)
Hemorrhage (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Obstructive shock (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischemia (Vascular disorders) | 0 (0) | 2 (2)
Shock (Vascular disorders) | 2 (2) | 3 (3)
Shock hemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mediastinal hematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mediastinal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary necrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 11 (11)
Thoracic hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 (3) | 4 (4)
Intestinal ischemia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Ischemic hepatitis (Hepatobiliary disorders) | 0 (0) | 4 (4)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Skin discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 10 (10)
Renal failure (Renal and urinary disorders) | 0 (0) | 4 (4)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Scrotum erosion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Catheter site thrombosis (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) — The cause of death of the participant was unknown. The SAE 'death' had the reported AE term 'Death not otherwise specified (NOS)'.
Generalised edema (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 3 (3) | 3 (3)
Edema peripheral (General disorders) | 0 (0) | 1 (1)
Prosthetic cardiac valve thrombosis (General disorders) | 1 (1) | 2 (2)
Vessel puncture site thrombosis (General disorders) | 1 (1) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dilutional coagulopathy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Graft hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 7 (7)
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural shock (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transfusion-related circulatory overload (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic hemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Venous injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Device pacing issue (Product Issues) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octaplex (N=213) | Frozen Plasma (N=207)
Bronchitis (Infections and infestations) | 1 (1) | 4 (4)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 3 (3)
Localised infection (Infections and infestations) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 4 (4)
Pneumonia (Infections and infestations) | 2 (2) | 6 (6)
Pneumonia klebsiella (Infections and infestations) | 2 (2) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 2 (2) | 4 (4)
Septic shock (Infections and infestations) | 4 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 5 (5)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 1 (1)
Wound infection (Infections and infestations) | 3 (3) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 65 (65) | 66 (66)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 3 (4) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 5 (5) | 4 (4)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (10) | 7 (8)
Hypersensitivity (Immune system disorders) | 3 (3) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Alkalosis hypochloremic (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (14) | 12 (12)
Hyperkalemia (Metabolism and nutrition disorders) | 9 (9) | 6 (6)
Hypervolemia (Metabolism and nutrition disorders) | 39 (39) | 42 (42)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 9 (11) | 15 (15)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (9) | 3 (3)
Hypovolemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Agitation (Psychiatric disorders) | 1 (2) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (3)
Confusional state (Psychiatric disorders) | 3 (3) | 2 (2)
Delirium (Psychiatric disorders) | 16 (16) | 14 (14)
Hallucination, visual (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 5 (6)
Altered state of consciousness (Nervous system disorders) | 2 (2) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 5 (5)
Cognitive disorder (Nervous system disorders) | 2 (2) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 2 (3)
ICU acquired weakness (Nervous system disorders) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Nystagmus (Nervous system disorders) | 2 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 6 (6)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Accelerated idioventricular rhythm (Cardiac disorders) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2) | 6 (6)
Atrial fibrillation (Cardiac disorders) | 87 (93) | 64 (68)
Atrial flutter (Cardiac disorders) | 11 (11) | 6 (7)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Atrioventricular block (Cardiac disorders) | 4 (4) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 9 (9) | 3 (3)
Atrioventricular block first degree (Cardiac disorders) | 3 (3) | 4 (4)
Atrioventricular block second degree (Cardiac disorders) | 3 (3) | 3 (3)
Bradycardia (Cardiac disorders) | 6 (6) | 3 (3)
Bundle branch block left (Cardiac disorders) | 4 (4) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 2 (2) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 5 (5)
Cardiac tamponade (Cardiac disorders) | 8 (8) | 5 (5)
Cardiogenic shock (Cardiac disorders) | 3 (3) | 8 (8)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 3 (3)
Nodal rhythm (Cardiac disorders) | 5 (5) | 6 (6)
Pericardial effusion (Cardiac disorders) | 4 (4) | 8 (8)
Pericarditis (Cardiac disorders) | 11 (11) | 7 (8)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 3 (3) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 4 (4) | 7 (7)
Supraventricular extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 2 (2)
Tachycardia (Cardiac disorders) | 7 (7) | 4 (4)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 4 (4) | 7 (7)
Deep vein thrombosis (Vascular disorders) | 4 (5) | 2 (2)
Distributive shock (Vascular disorders) | 2 (2) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (1) | 1 (1)
Hematoma (Vascular disorders) | 2 (2) | 3 (3)
Hemorrhage (Vascular disorders) | 5 (5) | 5 (5)
Hypertension (Vascular disorders) | 5 (5) | 4 (4)
Hypotension (Vascular disorders) | 17 (18) | 26 (27)
Peripheral ischemia (Vascular disorders) | 0 (0) | 3 (3)
Phlebitis (Vascular disorders) | 0 (0) | 3 (3)
Shock (Vascular disorders) | 2 (2) | 3 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 11 (12)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (9)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 28 (29) | 42 (44)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 28 (30) | 8 (8)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Rales (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 15 (15)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Thoracic hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 6 (6)
Dysphagia (Gastrointestinal disorders) | 5 (5) | 6 (6)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 (3) | 4 (4)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal ischemia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 23 (23) | 15 (15)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hypertransaminasemia (Hepatobiliary disorders) | 0 (0) | 2 (2)
Ischemic hepatitis (Hepatobiliary disorders) | 0 (0) | 4 (4)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 21 (21) | 36 (36)
Hematuria (Renal and urinary disorders) | 3 (3) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 4 (4)
Urinary retention (Renal and urinary disorders) | 4 (4) | 3 (3)
Chest pain (General disorders) | 5 (5) | 3 (3)
Chills (General disorders) | 2 (2) | 4 (4)
Generalised edema (General disorders) | 1 (2) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 3 (3) | 3 (3)
Edema (General disorders) | 2 (2) | 1 (1)
Edema peripheral (General disorders) | 33 (33) | 28 (28)
Prosthetic cardiac valve thrombosis (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 4 (4) | 3 (3)
Activated partial thromboplastin time prolonged (Investigations) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 2 (2)
Blood creatinine increased (Investigations) | 9 (9) | 4 (4)
Blood lactic acid increased (Investigations) | 0 (0) | 2 (2)
Blood potassium decreased (Investigations) | 1 (1) | 1 (1)
Breath sounds abnormal (Investigations) | 7 (7) | 6 (6)
Chest X-ray abnormal (Investigations) | 4 (4) | 1 (3)
Coagulation factor increased (Investigations) | 0 (0) | 3 (3)
Ejection fraction decreased (Investigations) | 1 (1) | 1 (1)
Hemoglobin decreased (Investigations) | 16 (17) | 16 (16)
Heart rate increased (Investigations) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 4 (4)
INR increased (Investigations) | 3 (3) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 2 (2)
Oxygen saturation decreased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 3 (3)
Troponin increased (Investigations) | 0 (0) | 4 (4)
Urine output decreased (Investigations) | 2 (2) | 1 (1)
Venous oxygen saturation decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count increased (Investigations) | 4 (4) | 2 (2)
Anemia postoperative (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Incision site pain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 10 (10)
Postoperative delirium (Injury, poisoning and procedural complications) | 0 (0) | 7 (7)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 12 (12) | 11 (11)
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/97/NCT05523297/Prot_002.pdf
  • Statistical Analysis Plan (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT05523297/SAP_003.pdf